### The GlaxoSmithKline group of companies

| Division | : | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | : | Reporting and Analysis Plan (RAP) |

| Title | : | Reporting and Analysis Plan for a double blind (sponsor open) placebo-controlled, stratified, parallel group study to evaluate the efficacy and safety of repeat doses of GSK3772847 in participants with moderate to severe asthma with allergic fungal airway disease (AFAD). |
|---|---|---|
| <b>Compound Number</b> | : | GSK3772847 |
| <b>Effective Date</b> | : | 24-JAN-2020 |

## **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 207972 (Document Number: 2017N331706 04)
- This RAP is intended to describe the Efficacy, Safety, PK, PD and Biomarker outputs required for the study.
- This RAP will be provided to the study team members to convey the content of the Statistical Analysis Complete (SAC) deliverable.

### **RAP Author(s):**

| Author | | Date |
|-----------------|--------------------------------------------|-------------|
| PPD | | 26-Nov-2019 |
| Principal Stati | stician (Respiratory, Clinical Statistics) | 20-NOV-2019 |

Copyright 2020 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

# **RAP Team Review Confirmations** (Method: E-mail)

| Reviewer | Date |
|---|---|
| Clinical Investigation Lead, Clinical Development Manager (Respiratory, Clinical Development) | 26-Nov-2019 |
| PPD PPD | |
| Programmer, Principal Programmer (Respiratory, Clinical Programming) | 26-Nov-2019 |
| PPD | |
| Pharmacokinetics, Senior Director (Respiratory, Clinical Pharmacology Modelling and Simulation) | 02-Dec-2019 |
| PPD | |
| Medical Monitor, Clinical Development Physician (Respiratory, MDC Global Clinical) | |
| PPD | |
| Project Physician Lead, Director of Clinical Development (Respiratory, MDC Global Clinical) | 10-Dec-2019 |
| PPD | |
| Value Evidence and Outcomes, Director Patient Centred<br>Outcomes, (Respiratory, Value Evidence and Outcomes) | 26-Nov-2019 |
| PPD | |
| Value Evidence and Outcomes, Scientist, Patient Centred Outcomes, (Respiratory, Value Evidence and Outcomes) | 26-Nov-2019 |

# Clinical Statistics & Clinical Programming Line Approvals (Method: Pharma TMF eSignature)

| Approver | Date |
|---------------------------------------------------------------|-------------|
| Senior Statistics Director (Respiratory, Clinical Statistics) | 13-Jan-2020 |
| Programming Manger (Respiratory, Clinical Programming) | 24-Jan-2020 |

## **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| 1. | INTRO | ODUCTION | 5 |
| 2. | SLIMI | MARY OF KEY PROTOCOL INFORMATION | 5 |
| ۷. | 2.1. | Changes to the Protocol Defined Statistical Analysis Plan | |
| | 2.2. | Study Objective(s) and Endpoint(s) | 6 |
| | 2.3. | Study Design | |
| | 2.4. | Statistical Analyses | |
| ^ | | NED ANALYOFO | • |
| 3. | | NED ANALYSES | |
| | 3.1. | Final Analyses | 9 |
| 4. | ANAL | YSIS POPULATIONS | 9 |
| | 4.1. | Analysis Populations | |
| | 4.2. | Protocol Deviations | 10 |
| 5. | CONS | SIDERATIONS FOR DATA ANALYSES AND DATA HANDLING | |
| | CON\ | /ENTIONS | 11 |
| | 5.1. | Study Treatment & Sub-group Display Descriptors | 11 |
| | 5.2. | Baseline Definitions | 11 |
| | 5.3. | Multicentre Studies | |
| | 5.4. | Examination of Covariates, Other Strata and Subgroups | 12 |
| | 5.5. | Multiple Comparisons and Multiplicity | 12 |
| | 5.6. | Other Considerations for Data Analyses and Data Handling Conventions | 12 |
| | | Conventions | 13 |
| 6. | STUD | Y POPULATION ANALYSES | 14 |
| | 6.1. | Overview of Planned Study Population Analyses | 14 |
| | 6.2. | Disposition | 14 |
| | 6.3. | Medical Conditions | 14 |
| | 6.4. | Concomitant Medications | 15 |
| 7. | EFFIC | CACY ANALYSES | 16 |
| | 7.1. | Primary Efficacy Analyses | |
| | 7.2. | Secondary Efficacy Analyses | |
| 8. | SAFF | TY ANALYSES | 17 |
| ٠. | 8.1. | Adverse Events Analyses | |
| | 8.2. | Vital Signs, Electrocardiogram (ECG) and Holter | |
| | 8.3. | Clinical Chemistry, Haematology and Cardiac Markers | |
| | 8.4. | Antibodies | |
| | 8.5. | Clinical Laboratory Analyses | 17 |
| 9. | PΗΔΕ | RMACOKINETIC ANALYSES | 12 |
| ٥. | 9.1. | Secondary Pharmacokinetic Analyses | |
| 10. | | RMACODYNAMIC AND BIOMARKER ANALYSES | |
| | TU.T. | Secondary Pharmacodynamic Analyses | 18 |

## CONFIDENTIAL

| 20 | 70 | 70 |
|-------------|-----|----|
| <i>-</i> /U | 7.9 | 72 |

| 11. | REFER | ENCES | | 18 |
|---|---|---|---|---|
| 12 | APPFI | NDICES | | 19 |
| 12. | 12.1. | | x 1: Protocol Deviation Management and Definitions for Per | |
| | 12.1. | Protocol | Population | 19 |
| | 12.2. | Annendi | x 2: Schedule of Activities | 20 |
| | 12.2. | 12.2.1. | | 20 |
| | 12.3. | | x 3: Assessment Windows | |
| | 12.0. | 12.3.1. | | |
| | 12.4. | _ | x 4: Study Phases and Treatment Emergent Adverse | 20 |
| | | | | 27 |
| | | 12.4.1. | | |
| | | 12.4.2. | Study Phases for Concomitant Medication | |
| | | 12.4.3. | Treatment Emergent Flag for Adverse Events | |
| | 12.5. | _ | x 5: Data Display Standards & Handling Conventions | |
| | 12.0. | 12.5.1. | Reporting Process | 29 |
| | | 12.5.2. | Reporting Standards | |
| | 12.6. | _ | x 6: Derived and Transformed Data | |
| | | 12.6.1. | General | |
| | | 12.6.2. | Study Population | |
| | | 12.6.3. | Safety | |
| | 12.7. | | x 7: Reporting Standards for Missing Data | |
| | | 12.7.1. | Premature Withdrawals | |
| | | 12.7.2. | Handling of Missing Data | |
| | | | 12.7.2.1. Handling of Missing and Partial Dates | |
| | 12.8. | Appendi | x 8: Values of Potential Clinical Importance | |
| | 12.9. | | x 9: Abbreviations & Trade Marks | |
| | | 12.9.1. | Abbreviations | |
| | | 12.9.2. | Trademarks | 37 |
| | 12.10. | Appendi | x 10: List of Data Displays | |
| | | | Data Display Numbering | |
| | | 12.10.2. | Mock Example Shell Referencing | 38 |
| | | | Deliverables | |
| | | | Study Population Tables | |
| | | 12.10.5. | Efficacy Tables | 42 |
| | | | Safety Tables | |
| | | | Pharmacokinetic Tables | |
| | | | Pharmacodynamic and Biomarker Tables | |
| | | | ICH Listings | |
| | | | ).Non-ICH Listings | |

## 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Study Report for Protocol of study 207972 (GSK Document No.: 2017N331706 03).

| Revision Chronology | ': | |
|---|---|---|
| 2017N331706_00 | 01-SEP-2017 | Original |
| 2017N331706_01 | 05-FEB-2018 | Clarified that participants with severe asthma for whom it is felt oral corticosteroids are warranted are not eligible for this study. |
| | | Clarified the use of anti-fungal medication throughout the study. |
| | | Clarified the run-in and randomisation criteria sections. |
| | | Clarified the timing of contraceptive requirements for female participants. |
| | | Provided a definition for former smokers. |
| | | Removed the body temperature in the objectives and safety analyses and updated Section 9 to reflect that body temperature will be collected but only available in source documents. |
| | | Corrected formatting and typographical errors. |
| 2017N331706_02 | 26-JUL-2018 | Russia specific: To allow Russian Federation Sites to conduct the screening assessments over 2 separate visits. |
| 2017N331706_03 | 10-OCT-2018 | To include participants with severe asthma with AFAD treated with low dose oral corticosteroid who still demonstrate a lack of complete control as demonstrated by ACQ-5, FeNO and blood eosinophil levels. Also, a few clarifications were included. |
| 2017N331706_04 | 10-OCT-2018 | Russia specific: To include participants with severe asthma with AFAD treated with low dose oral corticosteroid who still demonstrate a lack of complete control as demonstrated by ACQ-5, FeNO and blood eosinophil levels. Also, a few clarifications were included. |

# 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

Changes from the originally planned statistical analysis specified in the protocol are outlined in Table 1.

Table 1 Changes to Protocol Defined Analysis Plan

| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Statistical Analysis Plan | Statistical Analysis Plan | Rationale for Changes |
| Primary and secondary endpoints | All endpoints to be summarised | Enrolment into the 207972 study |
| to be analysed. | only. | was terminated early due to the |

| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Statistical Analysis Plan | Statistical Analysis Plan | Rationale for Changes |
| | | feasibility of completing the |
| | | study in a timely manner, |
| | | resulting in insufficient subjects |
| | | for analysis to be performed. |
| An internal Safety Review | No iSRC analysis and only one | The study was unable to recruit |
| Committee (iSRC) was to review | final SAC analysis to be performed. | the 20 randomised subjects |
| safety data after the 20th | | required for the iSRC prior to |
| randomised subject received their | | termination. |
| first post-dose ECG/24hr Holter. | | |
| | | In addition, as recruitment was |
| A potential interim analysis, end of | | terminated early, and would not |
| treatment analysis and final SAC | | inform internal decision making, |
| analysis was due to be performed. | | there was no requirement to |
| | | report at multiple timepoints to |
| | | align with portfolio decisions. |
| Primary, secondary and | Primary and secondary endpoints | As there is insufficient data to |
| exploratory endpoints to be | only to be reported. | draw any conclusions on |
| reported. | | exploratory endpoints, and they |
| | | are not required for external |
| | | disclosure, no outputs will be |
| | | created. |

# 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| To evaluate the efficacy of 3 doses of GSK3772847 (administered every 4 weeks) compared with | Change from baseline (Week 0) in blood eosinophils over time |
| placebo in moderate to severe asthma participants with allergic fungal airway disease (AFAD) who are currently on Standard of Care (SoC) | Change from baseline (Week 0) in fractional exhaled nitric oxide (FeNO) over time |
| Secondary Objectives | Secondary Endpoints |
| To evaluate the serum pharmacokinetics (PK) of 3 doses of GSK3772847 (administered every 4 weeks) in moderate to severe asthma participants with AFAD | Serum concentrations of GSK3772847 |
| To evaluate the pharmacodynamics (PD) of GSK3772847 in moderate to severe asthma participants with AFAD | Serum levels of free and total soluble suppressor of tumorigenicity 2 (sST2) |
| To evaluate the levels and specificity of any anti-<br>drug antibodies formed following dosing with<br>GSK3772847 | Incidence and titres of serum anti- GSK3772847 antibodies |
| To evaluate the health status of moderate to severe asthma participants with AFAD currently on SoC, and who are treated with GSK3772847 compared | Change from baseline (Week 0) in Asthma Control<br>Questionnaire -5 (ACQ-5) absolute score at Weeks 2, 4,<br>8 and 12 |
| with placebo-treated participants | Change from baseline (Week 0) in Asthma Quality of<br>Life Questionnaire (AQLQ) total and domain scores at<br>Weeks 2, 4, 8 and 12 |
| | Proportion of responders to ACQ-5. A responder to |

| Objectives | Endpoints |
|---|---|
| | ACQ-5 will be defined as a subject who has a decrease from baseline in ACQ-5 score of 0.5 or more at Weeks 2, 4, 8 and 12. • Proportion of responders to AQLQ. A responder to AQLQ will be defined as a subject who has an increase from baseline in AQLQ score of 0.5 or more at Weeks 2, 4, 8 and 12. |
| To evaluate the effect on lung function of moderate to severe asthma participants with AFAD currently on SoC, treated with GSK3772847 compared with placebo | Change from baseline (Week 0) in spirometry parameters over time including but not limited to pre-bronchodilator Forced expiratory volume in 1 second (FEV1). |
| To evaluate the safety and tolerability of GSK3772847 compared with placebo in moderate to severe asthma participants with AFAD | <ul> <li>Safety and tolerability parameters include:</li> <li>Treatment emergent adverse events (AE)</li> <li>Clinical Laboratory safety data</li> <li>Vital signs (blood pressure, heart rate)</li> <li>12–Lead Electrocardiogram (ECG) monitoring</li> <li>24-hour Holter monitoring</li> </ul> |
| Exploratory Objectives | Exploratory Endpoints |
| To evaluate changes in exploratory biomarkers in the blood of moderate to severe asthma participants with AFAD who have been treated with GSK3772847 compared with placebo | Change over time in levels of serum total<br>Immunoglobulin E (IgE), fungal-specific IgE |
| To evaluate changes in IL-33 related and disease biology biomarkers in the sputum of moderate to severe asthma participants with AFAD who have been treated with GSK3772847 compared with placebo | <ul> <li>Difference from placebo in levels of sputum biomarkers including but not limited to interleukin (IL)-33, IL-13, IL-4, IL-5 and TNF- α</li> <li>Difference from placebo including but not limited to levels of sputum eosinophils</li> </ul> |

## 2.3. Study Design



# 2.4. Statistical Analyses

Due to the study being terminated early, there were insufficient subjects to enable the planned statistical analysis to be performed. As a result, all data will be summarised descriptively only.

## 3. PLANNED ANALYSES

## 3.1. Final Analyses

The final planned analyses will be performed after the completion of the following sequential steps:

- 1. All participants have completed the study as defined in the protocol
- 2. All required database cleaning activities have been completed and database release has been declared by Data Management.
- 3. All criteria for unblinding the randomisation codes have been met.
- 4. Randomisation codes have been distributed according to RandAll NG procedures.
- 5. Database freeze (DBF) has been declared by Data Management.

## 4. ANALYSIS POPULATIONS

# 4.1. Analysis Populations

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Enrolled | The All Subjects Enrolled (ASE) population will consist of all participants who sign the ICF. | <ul> <li>Study population</li> <li>Subjects by country and site ID</li> <li>Age ranges</li> <li>Screening/run-in status and reason for screening/run-in failure.</li> </ul> |
| Screened | The screened population will consist of all participants who sign the ICF, but who did not pass the screening/run-in criteria and therefore were not randomised. | Reasons for<br>screen/run-in<br>failure |
| Randomised | The randomised population will consist of all participants who were randomised. A participant who is recorded as a screen or run-in failure and also randomised will be considered to be randomised in error provided they have not performed any study assessments. | No formal analysis<br>will be performed<br>on this population |
| Modified Intent-<br>to-Treat | <ul> <li>The modified Intent-to-Treat (mITT) will consist of all randomised participants who take at least 1 dose of study treatment.</li> <li>Participants will be analysed according to the treatment they receive &gt;=50% of the time. If the participant receives 50% of each treatment they will be analysed according to the randomised treatment.</li> </ul> | <ul> <li>Study population</li> <li>Inclusion,<br/>exclusion and<br/>randomisation<br/>criteria deviations</li> <li>Participant<br/>disposition</li> <li>Efficacy</li> </ul> |

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Safety | This population will be the same as the Modified Intent-to-<br>Treat population. | Safety |
| Pharmacokinetic | The PK population will consist of all randomised participants who received at least one dose of study medication, and for whom at least one pharmacokinetic sample was obtained, analysed and was measurable. | • PK |

Refer to Appendix 10: List of Data Displays which details the population used for each display.

### 4.2. Protocol Deviations

Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan [Version 2 (19-JUN-2018) or higher].

- Data will be reviewed prior to unblinding and freezing the database, to ensure all important deviations are captured and categorised on the protocol deviations dataset.
- This dataset will be the basis for the summaries and listings of protocol deviations.

A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the eCRF.

Note: Inclusion and exclusion criteria deviations are always reported as important.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

# 5.1. Study Treatment & Sub-group Display Descriptors

| | Treatment Group Descriptions | | |
|---|---|---|---|
| RandAll NG Data Displays for Reporting | | | |
| Code | Description | Description | Order [1] |
| G | GSK3772847 10 mg/kg | GSK3772847 | 2 |
| Р | Placebo | Placebo | 1 |

#### NOTES:

[1] Order represents treatments being presented in TFL, as appropriate

Treatment comparisons will be displayed as follows using the descriptors as specified:

• GSK3772847 vs Placebo

## 5.2. Baseline Definitions

For all endpoints (except as noted in baseline definitions) the baseline value will be the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. If time is not collected, Day 1 assessments are assumed to be taken prior to first dose and used as baseline.

| Parameter | | dy Assessm<br>dered as Ba | Baseline Used in<br>Data Display | |
|---|---|---|---|---|
| | Screening | Run-in | Day 1<br>(Pre-Dose) | |
| Primary Endpoints | | | | |
| Fractional Exhaled Nitric Oxide (FeNO) | Х | | Х | Day 1 |
| Blood Eosinophils | Х | | Х | Day 1 |
| Other Patient Reported Outcomes | 3 | | | |
| AQLQ | | | Х | Day 1 |
| Asthma Control Questionnaire (ACQ-5) score | Х | | Х | Day 1 |
| Spirometry | | | | |
| Forced Expiratory Volume (FEV1) | Х | | Χ | Day 1 |
| Pharmacodynamics | | | | |
| Free and total sST2 (serum) | | | Х | Day 1 |

| Parameter | | dy Assessm<br>dered as Ba | Baseline Used in<br>Data Display | |
|---|---|---|---|---|
| | Screening | Run-in | Day 1<br>(Pre-Dose) | |
| Safety | | | | |
| Vital Signs | Х | Х | Х | Day 1 |
| 12-lead Electrocardiogram (ECG) measurements | Х | | Х | Day 1 |
| 24 hours Holter measurements | | Χ | Х | Day 1 |
| Clinical laboratory tests (haematology and chemistry) | Х | | Х | Day 1 |
| Immunogenicity: Anti-<br>GSK3772847 antibodies | | | Х | Day 1 |
| Biomarkers | | | | |
| Induced sputum biomarkers | | Х | Х | Run-in <sup>1</sup> |
| Exploratory serum markers (including IgE and Fungal-specific IgE) | Х | | Х | Day 1 |

#### NOTES:

- Unless otherwise stated, the mean of replicate assessments taken on the same day will be used as the value for that day.
- Baseline is taken at run-in. If the sputum taken at run-in is not viable then a sample is taken at Day 1 (Pre-Dose) and is used as baseline.

## 5.3. Multicentre Studies

In this multicentre global study, enrolment will be presented by investigative site and country.

# 5.4. Examination of Covariates, Other Strata and Subgroups

No analysis will be performed on this data due to low subject numbers.

# 5.5. Multiple Comparisons and Multiplicity

No adjustment for multiplicity is required for this study, as no analysis will be performed.

# 5.6. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:

| Section | Component |
|---------|----------------------------------------------------------------|
| 12.3 | Appendix 3: Assessment Windows |
| 12.4 | Appendix 4: Study Phases and Treatment Emergent Adverse Events |
| 12.5 | Appendix 5: Data Display Standards & Handling Conventions |
| 12.6 | Appendix 6: Derived and Transformed Data |
| 12.7 | Appendix 7: Reporting Standards for Missing Data |
| 12.8 | Appendix 8: Values of Potential Clinical Importance |

## 6. STUDY POPULATION ANALYSES

## 6.1. Overview of Planned Study Population Analyses

The study population summaries will be based on the modified intent to treat population (mITT), unless specified to be on the All Subjects Enrolled (ASE) population.

Study population summaries including subject's disposition, protocol deviations, demographic and baseline characteristics, prior and concomitant medications, exposure and treatment compliance will be based on GSK Core Data Standards. Details of the planned displays are presented in Appendix 10: List of Data Displays.

## 6.2. Disposition

The study populations summary will use the All Subjects Enrolled (ASE) population and show the number of subjects overall who were enrolled, the number of screen failures and the number with each reason for screen failure. It will also show the number of subjects who were randomised and who were in the mITT, Safety and PK populations.

For the mITT population, two tables will be produced showing reasons for withdrawal from study and reasons for withdrawal from treatment. These summaries will show the number and percentage of subjects who completed the treatment/study, who withdraw prematurely and who reported each primary and sub-reason for withdrawal.

### 6.3. Medical Conditions

The number and percentage of subjects reporting each current medical condition will be presented. This table will include a subheading of 'Cardiovascular Risk Factors,' which will summarise the information taken from the cardiac disorders page in the eCRF. All medical conditions must be summarised on this table regardless of frequency. This will be repeated for past medical conditions.

## 6.4. Concomitant Medications

Non-Asthma medications will be summarised by Anatomical-Therapeutic-Chemical (ATC) level 1 and ingredient. Asthma medications will be summarised by the latest version of the Respiratory Medication Class (RMC), and will be derived for each asthma concomitant medication. Multi-ingredient medications will be presented according to their combination ATC classification rather than the classifications of the ingredients.

Asthma and non-asthma medications will be listed together. A listing of the relationship between ATC Level 1, ingredient and verbatim text will be produced for non-asthma medications only.

## 7. EFFICACY ANALYSES

Due to low subject numbers no statistical analysis will be performed.

# 7.1. Primary Efficacy Analyses

## 7.1.1. Endpoints and Summary Measures

| Primary Endpoints | Summary Measure |
|---|---|
| Change from baseline (Week 0) in blood eosinophils over | Summary statistics (raw and change from |
| time | baseline) |
| Change from baseline (Week 0) in fractional exhaled | Summary statistics (raw and change from |
| nitric oxide over time | baseline) |

Primary efficacy summaries will be based on the mITT population and no intercurrent events will be considered.

# 7.2. Secondary Efficacy Analyses

## 7.2.1. Endpoint and Summary Measure

| Secondary Endpoints | Summary Measure |
|---|---|
| <ul> <li>Change from baseline (Week 0) in spirometry parameters over time including but not limited to pre-bronchodilator Forced expiratory volume in 1 second.</li> <li>Change from baseline (Week 0) in Asthma Control Questionnaire -5 absolute score at Weeks 2, 4, 8 and 12</li> <li>Change from baseline (Week 0) in Asthma Quality of Life Questionnaire total and domain scores at Weeks 2, 4, 8 and 12</li> </ul> | Summary statistics (raw and change from baseline) |
| <ul> <li>Proportion of responders to ACQ-5. A responder to ACQ-5 will be defined as a subject who has a decrease from baseline in ACQ-5 score of 0.5 or more at Weeks 2, 4, 8 and 12.</li> <li>Proportion of responders to AQLQ. A responder to AQLQ will be defined as a subject who has an increase from baseline in AQLQ score of 0.5 or more at Weeks 2, 4, 8 and 12.</li> </ul> | Number and percentage of responders |

Secondary efficacy summaries will be based on the mITT population and no intercurrent events will be considered.

## 8. SAFETY ANALYSES

The safety analyses will be based on the Safety population, unless otherwise specified. The details of the planned displays are provided in Appendix 10: List of Data Displays.

## 8.1. Adverse Events Analyses

Adverse events analyses including the analysis of adverse events (AEs) and Serious (SAEs) will be based on GSK Core Data Standards.

## 8.2. Vital Signs, Electrocardiogram (ECG) and Holter

Summary statistics for vital signs at baseline, Weeks 0, 4, 8, 12, and 24 will be produced along with change from baseline summaries for each post baseline timepoint. In addition, the change between post-dose and pre-dose vital signs measurements will be summarised at weeks 0, 4 and 8.

A summary of ECG findings along with a table that shows the maximum increase in QTcF values post-baseline relative to baseline category will be produced.

In addition a summary of Holter interpretations will be produced for participants with at least 16 hours of data, however all data will be listed.

# 8.3. Clinical Chemistry, Haematology and Cardiac Markers

A summary of worst case clinical chemistry results relative to the normal range post-baseline, will be produced. Similar tables will be created for haematology and cardiac markers.

#### 8.4. Antibodies

Summaries of the incidence of and titres of anti- GSK3772847 antibodies at weeks 0\*, 2, 4\*, 8\*, 12 and 24.

\* = Pre-dose only

# 8.5. Clinical Laboratory Analyses

Laboratory evaluations including the analyses of liver function tests will be based on GSK Core Data Standards.

### 9. PHARMACOKINETIC ANALYSES

Due to low subject numbers no statistical analysis will be performed.

## 9.1. Secondary Pharmacokinetic Analyses

Serum concentrations of GSK3772847 will be summarised by nominal time.

Pharmacokinetic summaries will be based on the Pharmacokinetic population, and no intercurrent events will be considered.

## 10. PHARMACODYNAMIC AND BIOMARKER ANALYSES

## 10.1. Secondary Pharmacodynamic Analyses

Summary statistics of raw and percentage change from baseline in free and total soluble ST2 levels (serum) will be produced.

Pharmacodynamics summaries will be based on the mITT population, and no intercurrent events will be considered.

#### 11. REFERENCES

GlaxoSmithKline Document Number 2017N331706\_04, Protocol Amendment 2: A double blind (sponsor open) placebo-controlled, stratified, parallel group study to evaluate the efficacy and safety of repeat doses of GSK3772847 in participants with moderate to severe asthma with allergic fungal airway disease (AFAD). [10/OCT/2018].

Charter for the Internal Safety Review Committee (iSRC): A double blind (sponsor open) placebo-controlled, stratified, parallel group study to evaluate the efficacy and safety of repeat doses of GSK3772847 in participants with moderate to severe asthma with allergic fungal airway disease (AFAD). [30/JAN/2018]

Protocol Deviation Management Plan Version 2 (19-JUN-2018) or higher.

Winthrop et al, 2015, Opportunistic infections and biologic therapies in immune-mediated inflammatory diseases: consensus recommendations for infection reporting during clinical trials and postmarketing surveillance, Annals of the Rheumatoid Arthritis Disease, doi: 10.1136/annrheumdis-2015-207841. Epub 2015 Sep 22

## 12. APPENDICES

# 12.1. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population

The full list of protocol deviations collected on the eCRF is in the Protocol Deviation Management Plan (PDMP). Please refer to this document for current guidance.

There is no per protocol population in this study.

# 12.2. Appendix 2: Schedule of Activities Protocol Defined Schedule of Events

# 12.2.1.

| Procedure | Screening<br>(±5days) | Run-in<br>(±5days) | | Freatme<br>sit wind | to a reference | 770 | End of Treatment / EW (±3days) | FU (±3days) | Notes |
|---|---|---|---|---|---|---|---|---|---|
| Visit | V1 | V2 | V3 | V4 | V5 | V6 | V7 | V8 | |
| Week | -4 | -2 | 0 | 2 | 4 | 8 | 12 | 24 | |
| Day | -28 | -14 | 1 | 15 | 29 | 57 | 85 | 169 | |
| Informed consent | Χ | | | | | | | | May be obtained prior to Screening. |
| Inclusion and exclusion criteria | Х | X | X | | | | | | Recheck clinical status before 1st dose of study medication. |
| Demography | X | | | | | | | | |
| Full physical examination | X | | | | | | | | To include height and weight |
| Medical/medication/<br>drug/alcohol/smoking history | Χ | | | | | | | | Including smoking history, substance abuse,<br>medical conditions and family history of<br>premature cardiovascular disease; asthma<br>disease duration and exacerbation history |
| Human immunodeficiency virus (HIV), Hepatitis B and C screening | Х | | | | | | | | If test otherwise performed within 3 months prior to first dose of study treatment, testing at screening is not required |
| Genetics | | • | | 20 | | | | | |
| Informed consent for<br>Pharmacogenetic blood sample | 3 | X | | | | | | | |

| Procedure | Screening<br>(±5days) | Run-in<br>(±5days) | | Freatme<br>sit wind | | - | End of Treatment / EW (±3days) | FU (±3days) | Notes |
|---|---|---|---|---|---|---|---|---|---|
| Visit | V1 | V2 | V3 | V4 | V5 | V6 | V7 | V8 | |
| Week | -4 | -2 | 0 | 2 | 4 | 8 | 12 | 24 | |
| Pharmacogenetic (PGx) blood sample | | | | | X | | | | PGx sample may be drawn any time from Visit 3 onwards, pre-dose. Informed consent must be obtained before collecting a sample. |
| Study Treatment and Questionnaire | es | | | | | | | | ** |
| Randomisation | | | X | | | | | | |
| Study treatment | | | X | | X | X | | | |
| Dispense diary card | | X | | | | | | | To be completed daily. |
| Diary card review | | | X | X | X | X | X | | |
| Collect diary card | | | | | | | X | | |
| Rescue medication dispensing | | X | X1 | X1 | X1 | X <sup>1</sup> | | | As needed |
| ACQ-5 | X | | X | Х | X | Х | Х | | Test to be performed before all other assessments |
| AQLQ | | | X | X | X | X | X | | Test to be performed immediately after ACQ-5 |
| Efficacy | | | | ! | | | , , | | |
| Haematology (including eosinophil count) | X | | X1 | Х | Х | Х | X | | 1. Pre-dose |
| FeNO | X | | X | X | X | X | X | | Test to be performed pre-dose |
| Spirometry | X | | X | X | X | X | X | | Test to be performed pre-dose |

| Procedure | Screening (±5days) | Run-in<br>(±5days) | | Freatme<br>sit wind | | 100 | End of Treatment / EW (±3days) | FU (±3days) | Notes |
|---|---|---|---|---|---|---|---|---|---|
| Visit | V1 | V2 | V3 | V4 | V5 | V6 | V7 | V8 | |
| Week | -4 | -2 | 0 | 2 | 4 | 8 | 12 | 24 | |
| Free and total sST2 (serum) | | | X1 | х | X <sup>2</sup> | X <sup>1</sup> | Х3 | X3 | Pre and Post Dose Pre Dose Anytime (± 5 days) Pre-dose samples: within 2 hours from the planned dosing time Post-dose samples as soon as possible after end of infusion but must be taken within 4 hours. |
| Total & fungal specific IgE | X1 | | Χ2 | X | Х | X | Х | | Fungal specific IgE only if no historical documented results available Pre-dose |

| Procedure | Screening<br>(±5days) | Run-in<br>(±5days) | | | nt Perio<br>ow ±3da | | End of Treatment / EW (±3days) | FU (±3days) | Notes |
|---|---|---|---|---|---|---|---|---|---|
| Visit | V1 | V2 | V3 | V4 | V5 | V6 | V7 | V8 | |
| Week | -4 | -2 | 0 | 2 | 4 | 8 | 12 | 24 | |
| Induced sputum sample for biomarkers | | X | X12 | | | | Х3 | | <ol> <li>If no viable sample is produced at V2, induction should be repeated pre dose at V3</li> <li>If a participant does not produce a viable baseline sputum sample at visit 2 or at visit 3, the participant will not need to undergo a sputum induction at the end of the treatment period.</li> <li>If no viable sample is produced, induction should be repeated after a minimum of 72 hrs but no later than 7 days after scheduled visit.</li> </ol> |

| Procedure | Screening<br>(±5days) | Run-in<br>(±5days) | 1000 | | nt Perio<br>ow ±3da | 100 | End of Treatment / EW (±3days) | FU (±3days) | Notes |
|---|---|---|---|---|---|---|---|---|---|
| Visit | V1 | V2 | V3 | V4 | V5 | V6 | V7 | V8 | |
| Week | -4 | -2 | 0 | 2 | 4 | 8 | 12 | 24 | |
| Pharmacokinetics | | - 0 | | ·<br>2 | | | | ·<br>: | 5% |
| Serum blood sample for PK | | | X1 | Х | X <sup>2</sup> | X3 | X <sup>4</sup> | X <sup>4</sup> | Post Dose Pre Dose Pre and Post Dose Anytime (± 5 days) Pre-dose samples: within 2 hours from the planned dosing time Post-dose samples as soon as possible after end of infusion but must be taken within 4 hours. |
| Safety | | | - | | | | | | 1 |
| Laboratory assessments | X12 | | X1,3 | X <sup>1</sup> | X1,3 | X <sup>1</sup> | X1,3 | X <sup>1</sup> | Clinical chemistry (includes liver chemistry) Routine urinalysis at screening (Visit 1) Cardiac markers Note: haematology assessments in efficacy section |
| Serum blood sample for immunogenicity | | | X1 | Х | X1 | X1 | X | X | 1. Pre Dose |

| Procedure | Screening<br>(±5days) | Run-in<br>(±5days) | | Freatme<br>sit wind | | - | End of Treatment / EW (±3days) | FU (±3days) | Notes |
|---|---|---|---|---|---|---|---|---|---|
| Visit | V1 | V2 | V3 | V4 | V5 | V6 | V7 | V8 | |
| Week | -4 | -2 | 0 | 2 | 4 | 8 | 12 | 24 | |
| Urine or serum pregnancy test (WOCBP only) | × | 1 | X | | Х | Х | Х | X | To be performed pre-dose during the treatment period 1. Serum pregnancy test required |
| 12-lead ECG | Х | | X1 | | X1 | X1 | Х | | Test to be performed pre-dose and post-<br>dose within 30 mins after end of infusion. |
| 24 hour Holter | | Х | X1 | | | | | | Holter monitor needs to be returned to the clinic at end of 24 hour recording (i.e. the next day). 1Place the Holter 30-60mins prior to dosing |
| Vital signs | X | Х | X1 | | X1 | X1 | X | X | Test to be performed prior to the 12-lead<br>ECG (pre-dose and post dose) |
| AE review | | | <b>←===</b> | ===== | ===== | ===== | ===== | ===> | |
| SAE review | X | Χ | <b>←=======</b> | | | ====== | ===> | At V1 and V2 collect only SAEs considered as related to study participation. | |
| Concomitant medication review | X | X | <b>←===</b> | ===== | ===== | ===== | | ===> | |

EW: Early Withdrawal. The list of assessments listed in this column should be completed for an early withdrawal visit.

# 12.3. Appendix 3: Assessment Windows

# 12.3.1. Definitions of Assessment Windows for Analyses

Nominal visits will be used and no windowing will be applied for analysis.

# 12.4. Appendix 4: Study Phases and Treatment Emergent Adverse Events

## 12.4.1. Study Phases

Assessments and events will be classified according to the time of occurrence relative to study treatment start date.

| Study Phase | Definition |
|---|---|
| Pre-Treatment | Date ≤ Study Treatment Start Date |
| On-Treatment | Study Treatment Start Date < Date ≤ Study Treatment Stop Date + 28 days |
| Post-Treatment | Date > Study Treatment Stop Date + 28 days |

Completion of study epochs will be defined as the following:

| Study Phase | Definition of Completion |
|---|---|
| Run-in | Randomised into study and received first dose of study treatment |
| Treatment | Completed Week 12 visit |
| Follow up | Completed 12 week follow-up period |

# 12.4.2. Study Phases for Concomitant Medication

| Study Phase | Definition Note: All programming should use start and end dates where available, CMSTRF and CMENRF are only to be used where dates are unavailable to help determine the correct study phase. |
|---|---|
| Pre-Treatment | <ul> <li>Conmed Start Date &lt; Study Treatment First Dose Date</li> <li>Conmed End Date &lt; Study Treatment First Dose Date</li> <li>CMSTRF = "BEFORE"</li> <li>Randomisation date is missing i.e. subject was not randomised</li> </ul> |
| On-Treatment | <ul> <li>Study Treatment First Dose Date &lt;= Conmed Start Date &lt;= Study Treatment Last Dose Date + 28</li> <li>Study Treatment First Dose Date &lt;= Conmed End Date &lt;= Study Treatment Last Dose Date + 28</li> <li>(Conmed Start Date &lt;= Study Treatment Last Dose Date + 28) and (Conmed End Date &gt;= Study Treatment First Dose Date)</li> <li>(Conmed Start Date &lt;= Study Treatment Last Dose Date + 28) and (CMENRF = "DURING/AFTER" or CMENRF = "AFTER" or CMSTRF = "DURING")</li> <li>(CMSTRF = "BEFORE" or CMSTRF = "DURING" or CMENRF = "DURING/AFTER") and (Conmed End Date &gt;= Study Treatment First Dose Date)</li> <li>(CMSTRF = "BEFORE" or CMSTRF = "DURING") and (CMENRF = "DURING/AFTER" or CMENRF = "AFTER")</li> <li>CMSTRF = "DURING"</li> <li>CMSTRF = "DURING"</li> </ul> |
| Post-Treatment | Conmed Start Date > Study Treatment Last Dose Date + 28 |

| Study Phase | Definition Note: All programming should use start and end dates where available, CMSTRF and CMENRF are only to be used where dates are unavailable to help determine the correct study phase. |
|---|---|
| | <ul> <li>Conmed End Date &gt; Study Treatment Last Dose Date + 28</li> <li>CMENRF = "AFTER"</li> <li>CMENRF = "DURING/AFTER"</li> </ul> |
| All phases | Conmed start date is missing and CMSTRF is missing and conmed end date is missing and CMENRF is missing |

### NOTES:

- The duration of a single concomitant medication can extend over multiple study phases
- Please refer to Appendix 7: Reporting Standards for Missing Data for handling of missing and partial dates for concomitant medication. Use the rules in this table if concomitant medication date is completely missing.

# 12.4.3. Treatment Emergent Flag for Adverse Events

| Flag | Definition |
|---|---|
| Treatment | If AE onset date is on or after treatment start date & on or before treatment stop date + |
| Emergent | 28 days. |
| | Study Treatment Start Date ≤ AE Start Date ≤ Study Treatment Stop Date + 28 days |

#### NOTES:

• If the study treatment stop date is missing then the AE will be considered to be On-Treatment.

# 12.5. Appendix 5: Data Display Standards & Handling Conventions

## 12.5.1. Reporting Process

| Software | |
|---|---|
| The currently supported versions of SAS software will be used. | |
| Reporting Area | Reporting Area |
| HARP Server | : uk1salx00175 |
| HARP Compound | : /arenv/arprod/gsk3772847/mid207972/ |
| final_01:This is where | the end of study analysis will take place. |
| Analysis Datasets | |
| Analysis datasets will be created according to CDISC standards | |
| Generation of RTF Files | |
| RTF files will be generated for all reporting efforts | |

## 12.5.2. Reporting Standards

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated (IDSL Standards Location: https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics
- Do not include subject level listings in the main body of the GSK Clinical Study Report. All subject level listings should be located in the modular appendices as ICH or non-ICH listings

#### Formats

- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days
    on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.

#### **Unscheduled Visits**

Unscheduled visits will only be included in summary tables as part of 'minimum/maximum post baseline'

## CONFIDENTIAL

| and 'minimum/ma | and 'minimum/maximum change from baseline' summary. |
|---|---|
| <ul> <li>Unscheduled visit</li> </ul> | ts will not be included in figures. |
| All unscheduled v | risits will be included in listings. |
| <b>Descriptive Summar</b> | Descriptive Summary Statistics |
| Continuous Data Refer to IDSL Statistical Principle 6.06.1 | |
| Categorical Data | Categorical Data N, n, frequency, % |
| Graphical Displays | |
| Refer to IDSL Sta | Refer to IDSL Statistical Principals 7.01 to 7.13. |

## 12.6. Appendix 6: Derived and Transformed Data

#### 12.6.1. General

#### **Multiple Measurements at One Analysis Time Point**

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- If there are two values within a time window (as per Section 12.3.1) the value closest to the target day
  for that window will be used. If values are the same distance from the target, then the mean will be
  taken.
- Participants having both High and Low values for Normal Ranges at any post-baseline visit for safety parameters will be counted in both the High and Low categories of "Any visit post-baseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

## **Study Day**

- Calculated as the number of days from First Dose Date:
  - Ref Date = Missing → Study Day = Missing
  - Ref Date < First Dose Date → Study Day = Ref Date First Dose Date</li>
  - Ref Data ≥ First Dose Date → Study Day = Ref Date (First Dose Date) + 1

## 12.6.2. Study Population

### Age

Date of birth will be set as 30-JUN-YYYY where YYYY is the year of birth taken from the CRF. For participants who attended a screening visit, age will be calculated at the screening visit date.

## **Body Mass Index (BMI)**

BMI = Weight (kg) / Height(m)<sup>2</sup>

## **Treatment Misallocations**

To allocate treatment, the number of doses of GSK3772847 and Placebo that were given will be calculated, and the subject will be assigned to whichever treatment has the higher number. The only exception will be when both treatments were given equally, in which case the subject will be assigned their randomised treatment.

#### **Extent of Exposure (Therapeutic Coverage)**

- IP is administered approximately every 4 weeks and each dose viewed as providing therapeutic coverage for 4 weeks (28 days).
- Number of days of exposure to study drug will be calculated based on the formula:
  - Duration of Exposure in Days = Study Treatment Last Dose Date (Study Treatment First Dose Date) + 29
- The only exception to this will be when a participant dies in which case
   Duration of Exposure in Days = Death Date (Study Treatment First Dose Date) + 1

#### 12.6.3. Safety

### Maximum/Minimum On-Treatment Definitions for Vital Signs Data

Maximum and Minimum on-treatment: Maximum and Minimum on-treatment value over all time-points (including scheduled and unscheduled assessments) will be presented.

#### **Adverse Events**

### **Adverse Events of Special Interest (AESI)**

Systemic Allergic/Hypersensitivity and Non-allergic Reactions:

- Hypersensitivity (SMQ) [narrow]
- Anaphylactic reaction (SMQ) [narrow]
- Angioedema (SMQ) [narrow]

#### Alterations in immune response (infections)

All infections and serious infections reported under the MedDRA system organ class of 'Infections and Infestations'. Specific events of interest are opportunistic infections with preferred terms matching identified/pre-determined terms based on a published list of pathogens and/or presentations of specific pathogens to be considered as opportunistic infections in the setting of biologic therapy [Winthrop et al, 2015].

#### Alterations in immune response (malignancies):

All neoplasms reported under the MedDRA system organ class of 'Neoplasms, benign, malignant and unspecified (including cysts and polyps)'. Specific events of interest are malignancies which will be identified through matching of collected preferred terms with those from the following:

### Sub-SMQs under the Malignancies SMQ:

- Malignant tumours sub-SMQ (narrow terms)
- Tumours of unspecified malignancy sub-SMQ (narrow terms)

#### Alterations in cardiovascular safety:

Cardiac disorders and serious cardiac disorders reported under the MedDRA system organ class of 'Cardiac Disorders'. Serious cardiac, vascular and thromboembolic (CVT) events, identified as all serious events classified under the MedDRA system organ classes of 'Cardiac Disorders' and of 'Vascular Disorders', and thromboembolic events identified through matching of collected preferred terms with those from the following:

#### Sub-SMQs under the Embolic and thrombotic events SMQ:

- Embolic and thrombotic events, arterial sub-SMQ (narrow terms)
- Embolic and thrombotic events, venous sub-SMQ (narrow terms)
- Embolic and thrombotic events, vessel type unspecified and mixed arterial and venous sub-SMQ (narrow terms)

#### Sub-SMQs under the Ischaemic Heart Disease SMQ

- Mvocardial infarction sub-SMQ (narrow terms)
- Other Ischaemic heart disease sub-SMQ (narrow terms)

#### Sub-SMQs under the Central Nervous System Vascular Disorders SMQ

- Ischaemic central nervous system vascular conditions sub-SMQ (narrow terms)
- Central nervous system vascular disorders, not specified as haemorrhagic or ischaemic sub-SMQ (narrow terms)
- Serious ischemic adverse events, a subset of the serious CVT events identified through matching of collected preferred terms with those from the following:

#### Local Injection Site Reactions

Local injection site reactions are identifying through preferred terms which had been selected by medical review of the MedDRA dictionary and are provided in a separate spreadsheet.

# 12.7. Appendix 7: Reporting Standards for Missing Data

# 12.7.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Subject study completion (i.e. as specified in the protocol) was defined as completing the 12-week treatment period and three month safety follow up.</li> <li>Withdrawn participants were not replaced in the study.</li> <li>All available data from participants who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified.</li> </ul> |

# 12.7.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument:</li> <li>These data will be indicated by the use of a "blank" in subject listing displays. Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be missing data and should be displayed as such.</li> </ul> |
| Analysis | All missing data will be handled according to estimand of interest as described within the main body of the RAP. |
| ACQ-5 | <ul> <li>If one of the five items in the ACQ-5 is missing then the response from the four remaining items will be interpolated (pro-rata) to gain the overall response for the participant.</li> <li>If more than one item is missing then the ACQ-5 will be considered missing.</li> </ul> |
| AQLQ | <ul> <li>The AQLQ contains 32 items in four domains: activity limitation (11 items), symptoms (12 items), emotional function (five items), and environmental stimuli (four items). For the overall score, there must be no more than three missing responses (and never more than one per domain). The symptom and activity domain scores can have up to one missing value per domain, but for the emotional function and environmental stimuli domain scores must have no missing responses.</li> <li>If there are missing values at a visit (for example visit 2) then data will be imputed using data from both this visit and the previous study visit (for example visit 1) as shown below: <ul> <li>Visit 1 (completed data): Total score = A</li> <li>Visit 2 imputed score: B/A x 2</li> </ul> </li> </ul> |

# 12.7.2.1. Handling of Missing and Partial Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |
| Adverse | The eCRF allows for the possibility of partial dates (i.e., only month and year) to be |

| Events | recorded for AE start and end dates; that is, the day of the month may be missing. In such a case, the following conventions will be applied for calculating the time to onset and the duration of the event: o Missing Start Day: First of the month will be used unless this is before the start date of study treatment; in this case the study treatment start date will be used and hence the event is considered On-treatment as per Appendix 4: Study Phases and Treatment Emergent Adverse Events. o Missing Stop Day: Last day of the month will be used, unless this is after the stop date of study treatment; in this case the study treatment stop date will be used. Completely missing start or end dates will remain missing, with no imputation applied. Consequently, time to onset and duration of such events will be missing. |
|---|---|
| Concomitant<br>Medications/<br>Medical<br>History | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention: <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> </li> <li>The recorded partial date will be displayed in listings.</li> </ul> |

# 12.8. Appendix 8: Values of Potential Clinical Importance

Values of potential clinical importance will not be used in this study, instead normal reference ranges of "Low", "Normal" and "High" will be used.

# 12.9. Appendix 9: Abbreviations & Trade Marks

# 12.9.1. Abbreviations

| Abbreviation | Description |
|---|---|
| ACQ-5 | Asthma Control Questionnaire |
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| AFAD | Allergic Fungal Airway Disease |
| AIC | Akaike's Information Criteria |
| AQLQ | Asthma Quality of Life Questionnaire |
| ASE | All Subjects Enrolled |
| A&R | Analysis and Reporting |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| CPMS | Clinical Pharmacology Modelling & Simulation |
| CRO | Contract Research Organisation |
| CS | Clinical Statistics |
| CSR | Clinical Study Report |
| CTR | Clinical Trial Register |
| CV <sub>b</sub> /CV <sub>w</sub> | Coefficient of Variation (Between) / Coefficient of Variation (Within) |
| DBF | Database Freeze |
| DBR | Database Release |
| DOB | Date of Birth |
| DP | Decimal Places |
| ECG | Electrocardiogram |
| eCRF | Electronic Case Record Form |
| EOS | Eosinophils |
| FeNO | Fractional Exhaled Oxide |
| FEV1 | Forced expiratory volume in 1 second |
| HARP | Harmonisation of Analysis and Reporting Program |
| IA | Interim Analysis |
| ICF | Informed Consent Form |
| ICH | International Conference on Harmonisation |
| IDMC | Independent Data Monitoring Committee |
| IDSL | Integrated Data Standards Library |
| IgE | Immunoglobulin E |
| IMMS | International Modules Management System |
| IP | Investigational Product |
| iSRC | Internal Safety Review Committee |
| ITT | Intent-To-Treat |
| GUI | Guidance |
| LOC | Last Observation Carries Forward |
| mITT | Modified Intent-To-Treat |
| MMRM | Mixed Model Repeated Measures |
| PCI | Potential Clinical Importance |
| Abbreviation | Description |
|--------------|--------------------------------------------------|
| PD | Pharmacodynamic |
| PDMP | Protocol Deviation Management Plan |
| PGx | Pharmacogenetic |
| PK | Pharmacokinetic |
| POC | Proof of Concept |
| PP | Per Protocol |
| QC | Quality Control |
| QTcF | Frederica's QT Interval Corrected for Heart Rate |
| QTcB | Bazett's QT Interval Corrected for Heart Rate |
| RAP | Reporting & Analysis Plan |
| RAMOS | Randomisation & Medication Ordering System |
| RTF | Rich Text Format |
| SAC | Statistical Analysis Complete |
| SAE | Serious Adverse Event |
| SDTM | Study Data Tabulation Model |
| SoC | Standard of Care |
| SOP | Standard Operation Procedure |
| ST2 | Suppressor of Tumorigenicity 2 |
| TA | Therapeutic Area |
| TFL | Tables, Figures & Listings |
| WOCBP | Woman of Child Bearing Potential |
| GSK | GlaxoSmithKline |

### 12.9.2. Trademarks

| Trademarks of the GlaxoSmithKline<br>Group of Companies |
|---------------------------------------------------------|
| None |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| SAS |

#### 12.10. Appendix 10: List of Data Displays

All displays (Tables, Figures & Listings) will use the term 'Subjects' instead of "Participants".

#### 12.10.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------------------------|------------|------------|
| Study Population | 1.1 to 1.n | 1.1 to 1.n |
| Efficacy | 2.1 to 2.n | 2.1 to 2.n |
| Safety | 3.1 to 3.n | 3.1 to 3.n |
| Pharmacokinetic | 4.1 to 4.n | 4.1 to 4.n |
| Population Pharmacokinetic (PopPK) | 5.1 to 5.n | 5.1 to 5.n |
| Pharmacodynamic and / or Biomarker | 6.1 to 6.n | 6.1 to 6.n |
| Pharmacokinetic / Pharmacodynamic | 7.1 to 7.n | 7.1 to 7.n |
| Section | List | ings |
| ICH Listings | 1 t | 0 X |
| Other Listings | y t | 0 Z |

#### 12.10.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required example mock-up displays provided in Appendix 10: List of Data Displays: Example Mock Shells for Data Displays.

| Section | Figure | Table | Listing |
|------------------------------------|----------|----------|----------|
| Study Population | POP_Fn | POP_Tn | POP_Ln |
| Efficacy | EFF_Fn | EFF_Tn | EFF_Ln |
| Safety | SAFE_Fn | SAFE_Tn | SAFE_Ln |
| Pharmacokinetic | PK_Fn | PK_Tn | PK_Ln |
| Population Pharmacokinetic (PopPK) | POPPK_Fn | POPPK_Tn | POPPK_Ln |
| Pharmacodynamic and / or Biomarker | PD_Fn | PD_Tn | PD_Ln |
| Pharmacokinetic / Pharmacodynamic | PKPD_Fn | PKPD_Tn | PK/PD_Ln |

#### NOTES:

Non-Standard displays are indicated in the 'IDSL / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

### 12.10.3. Deliverables

| Delivery | Description |
|----------|-------------------------------------|
| SAC | Final Statistical Analysis Complete |

# 12.10.4. Study Population Tables

| Study I | Population Tab | les | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Disposition | | | | |
| 1.01. | mITT | ES8 | Summary of Subject Status and Reason for Study Withdrawal | ICH E3, FDAAA, EudraCT | SAC |
| 1.02. | mITT | SD4 | Summary of Treatment Status and Reasons for Discontinuation of Study Treatment | ICH E3 | SAC |
| 1.03. | mITT | ES4 | Summary of Subject Disposition at Each Study Epoch | ICH E3 | SAC |
| 1.04. | ASE | ES6 | Summary of Screening/Run-in Status and Reasons for Screen/Run-in Failure | Journal Requirements | SAC |
| 1.05. | ASE | NS1 | Summary of Number of Subjects by Country and Site ID | EudraCT/Clinical Operations | SAC |
| 1.06. | mITT | NS1 | Summary of Number of Subjects by Country and Site ID | EudraCT/Clinical Operations | SAC |
| Protoc | ol Deviation | | | | |
| 1.07. | mITT | DV1 | Summary of Important Protocol Deviations | ICH E3 | SAC |
| 1.08. | mITT | IE1 | Summary of Inclusion/ Exclusion Deviations | ICH E3 | SAC |
| Popula | tion Analysed | | | | |
| 1.09. | Enrolled | SP1 | Summary of Study Populations | IDSL. Footnote on population summary table that Safety and mITT populations are the same. | SAC |
| Demog | raphic and Bas | eline Characteris | tics | | |
| 1.10. | mITT | DM1 | Summary of Demographic Characteristics | ICH E3, FDAAA, EudraCT | SAC |
| 1.11. | Enrolled | DM11 | Summary of Age Ranges | EudraCT | SAC |
| 1.12. | mITT | DM5 | Summary of Race and Racial Combinations | ICH E3, FDA, FDAAA, EudraCT | SAC |

| Study F | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Prior a | Prior and Concomitant Medications | | | | |
| 1.13. | mITT | | Summary of Anti-Fungal Medications at Screening | | SAC |
| 1.14. | mITT | MH4 | Summary of Current Medical Conditions | ICH E3 | SAC |
| 1.15. | mITT | MH4 | Summary of Past Medical Conditions | ICH E3 | SAC |
| 1.16. | mITT | POP_T01 | Summary of Disease Duration and Exacerbation History | | SAC |
| 1.17. | mITT | CM1 | Summary of On-treatment Concomitant Medications | ICH E3 | SAC |
| 1.18. | mITT | CM1 | Summary of On-treatment Asthma Concomitant Medications | ICH E3 | SAC |

# 12.10.5. Efficacy Tables

| Efficac | y: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Primar | y Efficacy: Bloc | od Eosinophils an | d FeNO | | <u> </u> |
| 2.01. | mITT | EX1 | Summary of Exposure to Study Treatment | ICH E3 | SAC |
| 2.02. | mITT | | Summary of Raw and Change from Baseline in Blood Eosinophils | | SAC |
| 2.03. | mITT | | Summary of Raw and Change from Baseline in FeNO | | SAC |
| Second | dary Efficacy: S | Spirometry | | | |
| 2.04. | mITT | | Summary of Raw and Change from Baseline in FEV <sub>1</sub> | | SAC |
| Second | dary Efficacy: P | Patient Reported C | Outcomes | | |
| 2.05. | mITT | | Summary of Raw and Change from Baseline in ACQ-5 Total Score | | SAC |
| 2.06. | mITT | | Summary of ACQ-5 Responders | | SAC |
| 2.07. | mITT | | Summary of Raw and Change from Baseline in AQLQ Total Score | | SAC |
| 2.08. | mITT | | Summary of AQLQ Responders | | SAC |

# 12.10.6. Safety Tables

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | e Events (AEs) | | | | |
| 3.01. | SAFF | SAFE_T01 | Overview of On-treatment Adverse Events During the Study | | SAC |
| 3.02. | SAFF | AE1 | Summary of All On-treatment Adverse Events by System Organ Class and Preferred Term | ICH E3 | SAC |
| 3.03. | SAFF | AE1 | Summary of All On-treatment Serious Adverse Events by<br>System Organ Class and Preferred Term | ICH E3 | SAC |
| 3.04. | SAFF | AE3 | Summary of All On-treatment Adverse Events by Overall Frequency | ICH E3, summarise by PT | SAC |
| Labora | tory: Chemistry | / | | | |
| 3.05. | SAFF | LB1 | Summary of Worst Case Chemistry Results Relative to Normal Range Post-Baseline Relative to Baseline | ICH E3 | SAC |
| Labora | tory: Hematolo | gy and Cardiac M | arkers | | · |
| 3.06. | SAFF | LB1 | Summary of Worst Case Hematology and Cardiac Markers<br>Results Relative to Normal Range Post-Baseline Relative to<br>Baseline | ICH E3 | SAC |

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| ECG an | d Holter | | | | |
| 3.07. | SAFF | EG1 | Summary of ECG Findings | IDSL | SAC |
| 3.08. | SAFF | EG11 | Summary of Maximum Increase in QTcF Values Post-Baseline Relative to Baseline by Category | IDSL | SAC |
| 3.09. | SAFF | HM1 | Summary of Holter Interpretations | IDSL | SAC |
| Vital Si | gns | | | | |
| 3.10. | SAFF | VS1 | Summary of Vital Signs | ICH E3 | SAC |
| 3.11. | SAFF | VS1 | Summary of Change from Baseline in Vital Signs | ICH E3 | SAC |
| 3.12. | SAFF | VS1 | Summary of Change from Pre-dose to Post-dose in Vital Signs | ICH E3 | SAC |

#### 12.10.7. Pharmacokinetic Tables

| Pharma | Pharmacokinetic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Second | ary: Pharmaco | kinetic | | | |
| 4.01. | PK | | Summary of GSK3772847 Serum Pharmacokinetic Concentration-Time Data (ug/ml) | | SAC |
| 4.02. | PK | | Summaries of the Incidence of and Titres of Anti-<br>GSK3772847 Antibodies | | SAC |

### 12.10.8. Pharmacodynamic and Biomarker Tables

| Pharmacodynamic and Biomarker: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Second | Secondary Pharmacodynamic: Free and Total SST2 | | | | |
| 6.01. | mITT | | Summary of Raw and Percentage Change from Baseline in Free Soluble ST2 concentration (ug/mL) (On-treatment) | | SAC |
| 6.02. | mITT | | Summary of Raw and Percentage Change from Baseline in Total Soluble ST2 concentration (ng/mL) (On-treatment) | | SAC |

# 12.10.9. ICH Listings

| ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Disposition | | | | |
| 1. | Screened | ES7 | Listing of Reasons for Screen and Run-in Failure | Journal Guidelines | SAC |
| 2. | mITT | ES2 / ES3 | Listing of Reasons for Study Withdrawal | ICH E3 | SAC |
| 3. | mITT | SD2/SD3 | Listing of Reasons for Study Treatment Discontinuation | ICH E3 | SAC |
| 4. | mITT | BL1 / BL2 | Listing of Participants for Whom the Treatment Blind was Broken | ICH E3 | SAC |
| 5. | mITT | TA1 / CP_RD1x | Listing of Randomised and Actual Treatments | IDSL | SAC |
| Protoc | ol Deviations | | | | |
| 6. | mITT | DV2 | Listing of Important Protocol Deviations | ICH E3 | SAC |
| 7. | mITT | IE3 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | ICH E3 | SAC |
| Popula | tions Analysed | | | | |
| 8. | mITT | SP3 | Listing of Participants Excluded from Any Population | ICH E3. | SAC |
| Demog | raphic and Bas | eline Characteris | tics | | |
| 9. | mITT | DM2 | Listing of Demographic Characteristics | ICH E3 | SAC |
| 10. | mITT | DM9 | Listing of Race | ICH E3 | SAC |

| ICH: Li | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Prior a | nd Concomitan | t Medications | | | |
| 11. | mITT | CP_CM3 | Listing of Concomitant Medications | IDSL | SAC |
| Exposi | ure and Treatmo | ent Compliance | | | |
| 12. | mITT | EX3 | Listing of Exposure Data | ICH E3 | SAC |
| Advers | e Events | | | | |
| 13. | SAFF | AE8 | Listing of All Adverse Events | ICH E3 | SAC |
| 14. | SAFF | AE7 | Listing of Subject Numbers for Individual Adverse Events | ICH E3 | SAC |
| 15. | SAFF | AE8 | Listing of Adverse Events Leading to Withdrawal from Study / Permanent Discontinuation of Study Treatment | ICH E3 | SAC |
| 16. | SAFF | AE2 | Listing of Relationship Between Adverse Event System Organ Classes, Preferred Terms, and Verbatim Text | IDSL | SAC |
| Serious | s and Other Sig | nificant Adverse | Events | | |
| 17. | SAFF | AE8 | Listing of Fatal Serious Adverse Events | ICH E3 | SAC |
| 18. | SAFF | AE8 | Listing of Non-Fatal Serious Adverse Events | ICH E3 | SAC |
| 19. | SAFF | AE14 | Listing of Reasons for Considering as a Serious Adverse Event | ICH E3 | SAC |
| 20. | SAFF | AE8 | Listing of Serious Adverse Events Leading to Withdrawal from Study / Permanent Discontinuation of Study Treatment | ICH E3 | SAC |
| 21. | SAFF | AE8 | Listing of Adverse Events of Special Interest | ICH E3 | SAC |
| Hepato | biliary (Liver) | | | | • |
| 22. | SAFF | MH2 | Listing of Medical Conditions for Participants with Liver Stopping Events | IDSL | SAC |
| 23. | SAFF | SU2 | Listing of Substance Use for Participants with Liver Stopping Events | IDSL | SAC |

| ICH: Lis | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| All Lab | oratory | | | | |
| 24. | SAFF | LB5 / LB6 | Listing of All Laboratory Data for Participants with Any Value Outside Normal Range | ICH E3 | SAC |
| 25. | SAFF | LB14 | Listing of Laboratory Data with Character Results | ICH E3 | SAC |
| ECG | | | | | |
| 26. | SAFF | EG5 | Listing of All ECG Findings for Participants with an Abnormal ECG Finding | IDSL | SAC |
| Holter | 1 | | | | |
| 27. | SAFF | MH6 | Listing of Holter R-on-T Beat Data | IDSL | SAC |
| 28. | SAFF | MH7 | Listing of Holter {Supraventricular} {Ventricular} Event Data | IDSL, Update title as appropriate based on data | SAC |
| 29. | SAFF | MH8 | Listing of Holter {Sustained} {Non-sustained} {Supraventricular} {Ventricular} Run | IDSL, Update title as appropriate based on data | SAC |
| 30. | SAFF | MH9 | Listing of Holter Atrial {Fibrillation} {Flutter} Data | IDSL, Update title as appropriate based on data | SAC |
| 31. | SAFF | MH10 | Listing of Holter Abnormalities | IDSL | SAC |
| Vital Si | gns | | | | |
| 32. | SAFF | VS4 | Listing of All Vital Signs Data | IDSL | SAC |
| Primar | y Endpoint Data | a: Blood Eosinoph | nils and FeNO | | |
| 33. | mITT | | Listing of Blood Eosinophils | | SAC |
| 34. | mITT | | Listing of FeNO | | SAC |

# 12.10.10. Non-ICH Listings

| Non-IC | Non-ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Liver E | vents: Note on | ly produced if the | re is a Liver Event | | |
| 35. | SAFF | Patient Profile | Listing of Liver Events | | SAC |
| 36. | SAFF | Patient Profile | Listing of Liver Event Information for RUCAM Score | | SAC |
| 37. | SAFF | Patient Profile | Listing of Liver Biopsy | | SAC |
| 38. | SAFF | Patient Profile | Listing of Liver Imaging Details | | SAC |
| Cardio | ascular Event | s: Note only produ | uced if there is a Cardiovascular Event | | |
| 39. | SAFF | Patient Profile | Listing of Myocardial infarction/unstable angina | | SAC |
| 40. | SAFF | Patient Profile | Listing of Congestive heart failure | | SAC |
| 41. | SAFF | Patient Profile | Listing of Arrhythmias | | SAC |
| 42. | SAFF | Patient Profile | Listing of Valvulopathy | | SAC |
| 43. | SAFF | Patient Profile | Listing of Pulmonary hypertension | | SAC |
| 44. | SAFF | Patient Profile | Listing of Cerebrovascular events/stroke and transient ischemic attack | | SAC |
| 45. | SAFF | Patient Profile | Listing of Peripheral arterial thromboembolism | | SAC |
| 46. | SAFF | Patient Profile | Listing of Deep venous thrombosis/pulmonary embolism | | SAC |
| 47. | SAFF | Patient Profile | Listing of Revascularisation | | SAC |
| 48. | SAFF | Patient Profile | Listing of Deaths | | SAC |